CLINICAL TRIAL: NCT07038291
Title: Factors Associated With Extubation Failure in Kanigara ICU (Intensive Care Unit) RSUPN Dr. Cipto Mangunkusumo
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, Head of Anesthesiology and Intensive Care Study Program, Indonesia University
Other Study IDs: IndonesiaUAnes1006
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Extubation Failure; Ventilated Patients
Keywords: Extubation failure; ICU; Ventilator

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation Failure: Patient with extubation failure
  Interventions: Other: Not applicable- observational study
- Successful Extubation: Patient with successful extubation
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Observational study without intervention

SUMMARY:
Extubation is the final stage after patients undergo weaning procedure from mechanical ventilation in the ICU. Extubation failure followed by reintubation is associated with worse patient outcomes, including prolonged length of stay, increased risk of pulmonary infections, need for tracheostomy, higher healthcare costs, and increased mortality. Careful evaluation of various risk factors for extubation failure must be considered, therefore the extubation readiness guideline or checklist is essential before making the decision to extubate. This study aimed to identify factors associated with extubation failure in Kanigara ICU patients. This was a case-control study using secondary data from medical records of ICU patients who underwent extubation between January 2021 until August 2024. Variables analyzed included Glasgow Coma Scale (GCS) score, Arterial Blood Gas (ABG) results, hemodynamics, ventilator settings, airway protection ability, fluid balance, and airway-related problems. Bivariate and multivariate using logistic regression analyses were conducted to identify factors associated with extubation failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years old or more were intubated in Kanigara ICU RSCM more than 24 hours

Exclusion Criteria:

* Dead or needed tracheostomy before extubation, or reintubated for surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were intubated in Kanigara ICU for more than 24 hours in January 2021 until August 2024
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Factors Associated with Extubation Failure analyzed using logistic regression analysis | From January 2021 to August 2025
  Factors assessed were GCS score, hemodynamics, fluid balance, BGA results, airway protection ability, and airway related problems. Data were taken from medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkategowda PM, Mahendrakar K, Rao SM, Mutkule DP, Shirodkar CG, Yogesh H. Laryngeal air column width ratio in predicting post extubation stridor. Indian J Crit Care Med. 2015 Mar;19(3):170-3. doi: 10.4103/0972-5229.152763. PMID 25810614
- [Background] Xie J, Cheng G, Zheng Z, Luo H, Ooi OC. To extubate or not to extubate: Risk factors for extubation failure and deterioration with further mechanical ventilation. J Card Surg. 2019 Oct;34(10):1004-1011. doi: 10.1111/jocs.14189. Epub 2019 Aug 2. PMID 31374585
- [Background] Hazarika A, Singla K, Patel G, Mahajan V, Kahlon S, Meena S. Does Arterial Blood Gas (ABG) Provide a Safety Net for Extubation in Surgical Patients? Cureus. 2023 Jan 9;15(1):e33561. doi: 10.7759/cureus.33561. eCollection 2023 Jan. PMID 36779148
- [Background] Mokhlesi B, Tulaimat A, Gluckman TJ, Wang Y, Evans AT, Corbridge TC. Predicting extubation failure after successful completion of a spontaneous breathing trial. Respir Care. 2007 Dec;52(12):1710-7. PMID 18028561
- [Background] Godet T, Chabanne R, Marin J, Kauffmann S, Futier E, Pereira B, Constantin JM. Extubation Failure in Brain-injured Patients: Risk Factors and Development of a Prediction Score in a Preliminary Prospective Cohort Study. Anesthesiology. 2017 Jan;126(1):104-114. doi: 10.1097/ALN.0000000000001379. PMID 27749290
- [Background] Coplin WM, Pierson DJ, Cooley KD, Newell DW, Rubenfeld GD. Implications of extubation delay in brain-injured patients meeting standard weaning criteria. Am J Respir Crit Care Med. 2000 May;161(5):1530-6. doi: 10.1164/ajrccm.161.5.9905102. PMID 10806150
- [Background] Tanaka A, Shimomura Y, Uchiyama A, Tokuhira N, Kitamura T, Iwata H, Hashimoto H, Ishigaki S, Enokidani Y, Yamashita T, Koyama Y, Iguchi N, Yoshida T, Fujino Y. Time definition of reintubation most relevant to patient outcomes in critically ill patients: a multicenter cohort study. Crit Care. 2023 Sep 30;27(1):378. doi: 10.1186/s13054-023-04668-3. PMID 37777790
- [Background] Al-Husinat L, Jouryyeh B, Rawashdeh A, Robba C, Silva PL, Rocco PRM, Battaglini D. The Role of Ultrasonography in the Process of Weaning from Mechanical Ventilation in Critically Ill Patients. Diagnostics (Basel). 2024 Feb 12;14(4):398. doi: 10.3390/diagnostics14040398. PMID 38396437
- [Background] Andreu MF, Bezzi MG, Dotta ME. Incidence of immediate postextubation complications in critically Ill adult patients. Heart Lung. 2020 Nov-Dec;49(6):774-778. doi: 10.1016/j.hrtlng.2020.09.016. Epub 2020 Sep 24. PMID 32979642
- [Background] Epstein SK. Decision to extubate. Intensive Care Med. 2002 May;28(5):535-46. doi: 10.1007/s00134-002-1268-8. Epub 2002 Apr 12. PMID 12029399
- [Background] Arcanjo ABB, Beccaria LM. Factors associated with extubation failure in an intensive care unit: a case-control study. Rev Lat Am Enfermagem. 2023;31:e3864. doi: 10.1590/1518-8345.6224.3864. PMID 36995853
- [Background] Kulkarni AP, Agarwal V. Extubation failure in intensive care unit: predictors and management. Indian J Crit Care Med. 2008 Jan;12(1):1-9. doi: 10.4103/0972-5229.40942. PMID 19826583
- See also: Related Info — https://www.ui.ac.id/akademik/fakultas/fakultas-kedokteran/